CLINICAL TRIAL: NCT06283342
Title: The Role of Prophylactic Iron Use and Nutrition in Preventing Iron Deficiency in Infancy
Brief Title: Prophylactic Iron and Nutrition in Preventing Infant Iron Deficiency
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, Principal Investigator, Konya Meram State Hospital
Other Study IDs: Konya Pediatric Hematology
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Iron Deficiency Anemia in Childbirth; Infant Nutrition Disorders; Iron Deficiencies
Keywords: prophylactic iron; infant nutrition; iron deficiency prevention; pediatric health
MeSH Terms: conditions — Infant Nutrition Disorders; Iron Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Iron deficiency group: Patients with a ferritin level below 12 mg/L were considered to have Iron deficiency group.
- Not iron deficiency group: Patients with a ferritin level above 12 mg/L were considered to have not iron deficiency group.
- Iron deficiency anemia group: Patients with ferritin level below 12 mg/L and hemoglobin (Hb) value below 11 g/dL were considered to have IDA.
- Not iron deficiency anemia group: Patients with ferritin level below 12 mg/L and hemoglobin (Hb) value above 11 g/dL were considered to have Not iron deficiency anemia group.

SUMMARY:
This study aimed to reveal the effects of prophylactic iron preparations, adequate breast milk intake, and iron-rich supplementary food intake in the prevention of IDA (iron deficiency anemia) and ID (iron deficiency) in infancy.

DETAILED DESCRIPTION:
Iron plays an important role in oxidation and reduction reactions, which have a very important place in the continuation of life. Iron plays an essential role in these reactions because it can easily gain and lose electrons in redox reactions. Iron is mostly found in the heme molecule in organisms. However, iron has structural and functional importance for many enzymes and proteins other than heme. Iron deficiency (ID) is the most common nutritional deficiency in children worldwide. ID is more common in socio-economically developing geographies. However, it is still an important problem in developed countries. A plasma ferritin level below 12 mg/L is defined as ID, which is often used synonymously with iron deficiency anemia (IDA). However, ID develops before anemia occurs. Weakness, fatigue, tiring quickly, insomnia, and regression in neuro-cognitive functions may occur in ID that precedes the signs of anemia. With the development of anemia, the clinical diagnosis of IDA is fully revealed.

In ID that occurs in infancy, psychomotor development is adversely affected, and the development of cognitive functions slows down or even stops. Immune system functions regress. Although iron treatment can reverse these negative effects, some effects are permanent. Therefore, prevention of ID is more important than treatment. In addition, it is easier and cheaper to prevent ID and IDA than to treat them. It is a health policy to recommend iron prophylaxis to children aged 4-12 months in the Republic of Turkey.

Adding iron-rich foods to the diet, adequate breast milk intake, and prophylaxis with iron preparations can be used to prevent ID and IDA. However, there are different data in the literature on the use of prophylactic iron preparations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 6-24 months and admitted to the general pediatrics outpatient clinic

Exclusion Criteria:

* Chronic disease
* Blood transfusion history,
* Thalassemia carrier status
* Clinical diagnosis of infection or elevated C-reactive protein (CRP)
* Patients who received iron deficiency or iron deficiency anemia treatment
* Those who were born prematurely
* Patients with low birth weight

Ages: 6 Months to 24 Months | Sex: All
Age Groups: Child
Gender Based: Yes — Patients aged between 6-24 months and admitted to the general pediatrics outpatient clinic were included in the study
Study Population: Study population include children aged 6-24 months, who were admitted to the general pediatric outpatient clinic of our hospital between January 1st, 2018, and February 1st, 2019.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Ferritine level | day 1
  Ferritin level below 12 mg/L was considered iron deficiency.

SECONDARY OUTCOMES:
Hemoglobin level | day 1
  Hemoglobin (Hb) values below 11 g/dL were considered as having anemia
Prophylactic iron use rate | 15 days
  Giving 10 mg/day iron drops to babies starting from the 4th month was considered as the correct prophylaxis recommendation. Prophylactic iron use rates were calculated by dividing those using iron prophylaxis in all groups by the number of participants in the groups.
Iron-sufficient supplementary food intake rate of babies | 15 days
  Babies whose mothers answered "yes" to at least two of the following questions in the survey evaluating babies' iron-sufficient supplementary food intake were considered to be fed adequately in terms of iron:
  * Does your baby eat 1 egg at least 3 days a week?
  * Does your baby eat meat the size of 2 meatballs 2 days a week?
  * Does your baby eat legumes at least 3 times a week? This ratio was calculated by dividing the number of adequately nourished participants by the total number of participants in the group.
Breast milk usage rate | 15 days
  Exclusive breastfeeding for at least 6 months after birth was considered adequate breast milk intake. Those who breastfed during this period were considered to have used sufficient breast milk. The breast milk usage rate was found by dividing those who received adequate breast milk by the participants in the group.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Derived] Simsek A, Energin VM. The role of prophylactic iron utilization and nutrition to prevent iron deficiency in infancy: Prospective cohort study. Medicine (Baltimore). 2025 Jun 13;104(24):e42947. doi: 10.1097/MD.0000000000042947. PMID 40527768